CLINICAL TRIAL: NCT07226479
Title: Non-invasive Central Venous Pressure Estimation in Cardiac Intensive Care
Brief Title: Non-invasive Venous Pressure Estimation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Compremium AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2000040660
Record Dates: First submitted 2025-11-06; First posted 2025-11-10 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Cardiac Intensive Care

STUDY DESIGN:
Intervention Model Description: Adult patients admitted to the CICU with invasive CVP/RA pressure measurements (Central line or pulmonary artery catheter) placed by standard of care as determined by the treating team before enrollment. With-in participant design.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Adult CICU patients- CPMX2 (Experimental): Adult participants admitted to the CICU will have external jugular venous occlusion pressure measured twice non-invasively with the venous occlusion pressure monitoring device (CPMX2) and twice using standard of care invasive central venous pressure (CVP) measurements. All measurements will be taken concurrently. This is a with-in participant design.
  Interventions: Device: CPMX2

INTERVENTIONS:
Device: CPMX2 — Non-invasive venous occlusion pressure monitoring device

SUMMARY:
The non-invasive central venous pressure estimation in adult cardiac intensive care units (CICU) patients study is a single-center, single-arm, investigator-blinded, interventional, intra-participant comparative, feasibility study. This study aims to assess the safety and preliminary accuracy of external jugular venous occlusion pressure measured non-invasively with the venous occlusion pressure monitoring device (CPMX2) in adult CICU patients. As a feasibility study, the primary goal is to gather preliminary data on the feasibility, safety, and effectiveness of the non-invasive CVP estimation method. Although single arm, the study will compare non-invasive CVP measurements with standard invasive CVP measurements taken concurrently. This intra-participant comparative approach is essential to validate the correlation and reliability of the non-invasive method.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent
* Admitted to the CICU with invasive CVP/RA pressure monitoring placed by standard of care as determined by the treating team before enrollment
* No more than moderate TR as assessed by echocardiogram

Exclusion Criteria:

* Undergoing positive pressure ventilation (Bipap or invasive mechanical ventilation)
* Non-visible external jugular vein bilaterally (by visual examination or with traditional ultrasound examination)
* History of thrombosis in any of the following vessels bilaterally; external jugular vein, internal jugular vein, brachiocephalic vein or superior vena cava
* Skin lesions, vascular access sites or dressings covering neck and impeding access to the external jugular veins at the level of the muscle belly of the sternocleidomastoid muscle

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-06 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Mean venous pressure to assess accuracy | Day 1
  Mean CPMX2 external jugular occlusion pressure will be compared to invasive CVP measurement in mmHg
Number of adverse events to assess safety | Day 1
  Safety measured by number of adverse events related to or potentially related to the study device and device deficiencies reported during study
Number of device deficiencies to assess safety | Day 1
  Safety measured by number of device deficiencies reported during study

SECONDARY OUTCOMES:
Mean Point-of-care ultrasound (POCUS)-derived pressure measurements | Day 1
  Mean POCUS-derived pressure measurements as defined by current clinical guidelines (calculated using inferior vena cava (IVC) collapsibility and diameter measurements)

CONTACTS AND LOCATIONS:
Overall Officials: Elliott Miller, MD, MHS, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital CICU, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No